CLINICAL TRIAL: NCT05470348
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of BL-B01D1 in Patients With Unresectable Locally Advanced or Metastatic Breast Cancer and Other Solid Tumors
Brief Title: A Study of BL-B01D1 in Patients With Unresectable Locally Advanced or Metastatic Breast Cancer and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry); Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-104
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Solid Tumor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1 (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507

SUMMARY:
In this study, the dose-limiting toxicity (DLT), maximum tolerated dose (MTD), recommended phase II dose (RP2D), the preliminary efficacy, pharmacokinetic characteristics, and immunogenicity of BL-B01D1 will be investigated in patients with unresectable locally advanced or metastatic breast cancer and other solid tumors.

DETAILED DESCRIPTION:
In phase Ia, the safety and tolerability of BL-B01D1 in patients with unresectable locally advanced or metastatic breast cancer and other solid tumors. investigated to determine the dose-limiting toxicity (DLT), and maximum tolerated dose (MTD) of BL-B01D1.

In phase Ib, the safety and tolerability of BL-B01D1 at the phase Ia recommended dose will be further investigated, and recommended phase II dose (RP2D) for phase II clinical studies will be determined The preliminary efficacy, pharmacokinetic characteristics, and immunogenicity of BL-B01D1 in patients with locally advanced or metastatic solid tumors will be evaluated.

EGFR and/or HER3 protein expression or gene amplification in tumor pathological tissues will be detected, and the expression of related ligand will be explored to study its correlation with the validity index of BL-B01D1, and the biomarkers will be optimized to further study the correlation between selected biomarkers and initial efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. No gender restrictions;
3. Age: ≥18 years and ≤75 years;
4. Expected survival time ≥3 months;
5. Histologically and/or cytologically confirmed unresectable locally advanced or metastatic breast cancer and other solid tumors with failed standard treatment, intolerance to standard treatment, no current standard treatment available, or inability to access standard treatment;
6. Enrolled subjects should not have received prior systemic therapy for unresectable locally advanced or recurrent/metastatic triple-negative breast cancer;
7. Agree to provide archived tumor tissue specimens or fresh tissue samples from primary or metastatic lesions within the past 3 years;
8. Must have at least one measurable lesion as defined by RECIST v1.1;
9. ECOG performance status score of 0 or 1;
10. Toxicity from prior anti-tumor therapy has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
11. No severe cardiac dysfunction, with left ventricular ejection fraction (LVEF) ≥50%;
12. Organ function levels must meet the requirements without transfusion or use of any cell growth factors and/or platelet-raising drugs within 14 days before the first dose of the study drug;
13. Coagulation function: International Normalized Ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5 × ULN;
14. Urine protein ≤2+ or ≤1000 mg/24h;
15. For premenopausal women with childbearing potential, a pregnancy test (serum or urine) must be performed within 7 days before starting treatment, and the result must be negative; they must not be breastfeeding. All enrolled patients (regardless of gender) must use adequate barrier contraception throughout the treatment period and for 6 months after treatment ends.

Exclusion Criteria:

1. Received biological therapy, immunotherapy, or other antitumor treatments within 4 weeks or 5 half-lives prior to the first dose (6 weeks for mitomycin and nitrosoureas; oral fluorouracil drugs such as tegafur/gimeracil/oteracil (S-1) or capecitabine, or oral endocrine therapy, or palliative radiotherapy within 2 weeks before the first dose);
2. History of severe heart disease;
3. Prolonged QT interval, complete left bundle branch block, third-degree atrioventricular block, or severe arrhythmia;
4. Active autoimmune or inflammatory diseases;
5. Diagnosis of other malignancies within 2 years prior to the first dose;
6. Poorly controlled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg) despite the use of two antihypertensive medications;
7. Poorly controlled blood glucose (defined as: a) two fasting blood glucose levels >10 mmol/L, or b) glycated hemoglobin level exceeding 8%), or concurrent diabetic gangrene;
8. History of interstitial lung disease (ILD), current ILD, or suspected ILD based on imaging during screening;
9. Concurrent pulmonary disease leading to clinically significant respiratory impairment;
10. Unstable deep vein thrombosis, arterial thrombosis, pulmonary embolism, or other thrombotic events requiring therapeutic intervention within 6 months before screening (excluding catheter-related thrombosis);
11. Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (leptomeningeal metastases);
12. Patients with significant serous cavity effusion, symptomatic effusion, or poorly controlled effusion;
13. History of hypersensitivity to recombinant humanized antibodies or human-mouse chimeric antibodies, or any excipients of BL-B01D1;
14. Imaging findings indicating tumor invasion or encasement of major thoracic, cervical, or pharyngeal blood vessels, unless the investigator deems it does not affect the patient's eligibility for treatment;
15. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
16. Cumulative anthracycline dose >360 mg/m² in prior (neo)adjuvant anthracycline therapy;
17. Positive for human immunodeficiency virus antibody (HIVAb), active tuberculosis, active hepatitis B virus (HBV) infection, or active hepatitis C virus (HCV) infection;
18. Severe infection (CTCAE > Grade 2) within 4 weeks before the first dose of the study drug; signs of active pulmonary infection within 2 weeks before the first dose;
19. Participation in another clinical trial within 4 weeks before the first dose (calculated from the last dose date);
20. Any other condition deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ib: phase II clinical studies (RP2D) | Up to 21 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.
Phase Ia: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  In the dose escalation stage, MTD was selected as the highest dose whose DLT rate estimate was closest to the target DLT rate, but did not exceed the upper bound of the EQUIVALENT interval of DLT rate.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1 . The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1 .
Cmax | Up to 21 days after the first dose
  Maximum serum concentration (Cmax) of BL-B01D1 will be investigated
Tmax | Up to 21 days after the first dose
  Time to maximum serum concentration (Tmax) of BL-B01D1 will be investigated
T1/2 | Up to 21 days after the first dose
  Half-life (T1/2) of BL-B01D1 will be investigated
AUC0-t | Up to 21 days after the first dose
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration
Ctrough | Up to 21 days after the first dose
  Ctough is defined as the lowest serum concentration of BL-B01D1 prior to the next dose will be administered
ADA (anti-drug antibody） | Up to approximately 24 months
  The anti-drug antibody of BL-B01D1
Nab (neutralizing antibody) | Up to approximately 24 months
  Neutralizing anti-drug antibodies produced by BL-B01D1
Objective Response Rate（ORR） | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Progression-free Survival(PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-B01D1 to the first date of either disease progression or death, whichever occurs first.
CL (Clearance) | Up to approximately 24 months
  CL in the serum of BL-B01D1 per unit of time will be investigated

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, Principal Investigator — Fudan University; Jian Zhang, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Fudan University ShangHai Cancer Center, Shanghai, Shanghai Municipality